CLINICAL TRIAL: NCT02786277
Title: Uplift Modeling to More Narrowly Target Alerts for Acute Kidney Injury
Brief Title: Learning Alerts for Acute Kidney Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YALEAKIALERTLEARN; 1R01DK113191-01A1 (NIH)
Record Dates: First submitted 2016-05-13; First posted 2016-05-30 (Estimated); Results first posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recommended (Experimental): Those whose uplift score represents a probability of benefit greater than 0.5 will generate an alert, while those whose uplift score represents a probability of benefit less than 0.5 will not generate an alert.
  Interventions: Other: Alert
- Anti-recommended (Experimental): Those whose uplift score represents a probability of benefit greater than 0.5 will not generate an alert, while those whose uplift score represents a probability of benefit less than 0.5 will generate an alert.
  Interventions: Other: Alert

INTERVENTIONS:
Other: Alert — An alert informing the provider of the presence of acute kidney injury will be fired.

SUMMARY:
The primary objective of this study is to determine whether the use of uplift (also known as Conditional Average Treatment Effect - CATE) modeling to empirically identify patients expected to benefit the most from AKI alerting and to target AKI alerts to these patients will reduce the rates of AKI progression, dialysis, and mortality.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) carries a significant, independent risk of mortality among hospitalized patients, but despite its association with poor clinical outcomes, AKI is asymptomatic and frequently overlooked by clinicians, with fewer than half of all AKI patients with documentation of the syndrome in the electronic medical record, which was associated with decreased rates of AKI clinical best practices.

Our research group recently conducted a large-scale multicenter randomized controlled trial of electronic alerts for AKI throughout the Yale New Haven Health System from 2018 to 2020 (ELAIA-1). Our study showed that, overall, alerting physicians to the presence of AKI did not demonstrate a difference in the rate of our primary outcome of progression of AKI, dialysis, or death, despite the alert leading to some process of care changes such as measurement of creatinine and urinalysis. There was, however, substantial heterogeneity among the study sites. The proliferation of alerting systems that are ineffective can lead to the phenomenon of alert fatigue, whereby providers tend to ignore alerts in a high-alert environment, and can have deleterious effects on patient care. Further, given the highly heterogenous nature of AKI, a more personalized approach to AKI alerting may be warranted.

Uplift modeling, commonly used in marketing, is a novel concept in the medical field and aims to determine phenotypic characteristics that predict a response (benefit or harm) to a given intervention. In this way, patients who are predicted to benefit most from an intervention are identified and preferentially targeted. Uplift modeling of alerting systems has the potential to both improve alert effectiveness through intelligent targeting, and reduce alert fatigue.

In this study, we will expand upon our prior AKI alert trial to determine prospectively whether the use of uplift modeling to preferentially target patients expected to benefit from an AKI alert will reduce the rates of AKI progression, dialysis and death among hospitalized patients with AKI. Inpatients at 4 teaching hospitals within the YNHH system with AKI, based on the Kidney Disease: Improving Global Outcomes (KDIGO) creatinine criteria, will be randomized to a "recommended" group (with higher scores receiving alerts and lower scores not receiving alerts as recommended) versus an "anti-recommended" group (with higher scores not receiving alerts and lower scores receiving alerts as anti-recommended). The primary outcome will be a composite of AKI progression, dialysis, or mortality within 14 days of randomization. Secondary outcomes will focus on AKI-specific process measures.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years
2. Admitted to a participating hospital
3. Has AKI as defined by creatinine criteria:

   * 0.3 mg/dl increase in inpatient serum creatinine over 48 hours OR
   * 50% relative increase in inpatient serum creatinine over 7 days

Exclusion Criteria:

1. Dialysis order prior to AKI onset
2. Initial creatinine ≥ 4.0 mg/dl
3. Prior admission in which patient was randomized
4. Admission to hospice service or comfort measures only order
5. ESKD diagnosis code
6. Kidney transplant within six months
7. Opted out of electronic health record research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2046 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2025-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis P Wilson, MD MSCE, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data underlying results for publication will be made available upon publication of results.
Supporting Information: Study Protocol, SAP
Time Frame: Upon publication of results; indefinitely

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred at 4 hospital sites across the Yale New Haven Hospital System. Identification of eligible patient subjects was performed within the Epic electronic medical record system based on inclusion and exclusion criteria by an algorithm embedded into the best practice alert. Randomization occurred the moment the best practice build identified a patient as being eligible.
Period: Overall Study
Arm/Group | Recommended | Anti-recommended
Started | 1002 | 1044
Completed | 1002 | 1044
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Recommended | Anti-recommended | Total
Number analyzed (Participants) | 1002 | 1044 | 2046
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 64.5 [41 to 74.1] | 63.2 [34.1 to 73.9] | 63.7 [36.6 to 74]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 537 | 503 | 1040
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 188 | 206 | 394
  Hispanic or Latino | 108 | 140 | 248
Creatinine mg/dL [Median (Inter-Quartile Range); unit: mg/dL] | 1.5 [1.1 to 2] | 1.5 [1.1 to 2] | 1.5 [1.1 to 2]
Diastolic blood pressure (mmHg) [Median (Inter-Quartile Range); unit: mmHg] | 67 [60 to 76] | 68 [61 to 77] | 68 [60 to 76]
Pulse (bpm) [Median (Inter-Quartile Range); unit: beats per minute] | 80 [69 to 93] | 80 [69 to 91.8] | 80 [69 to 92]
Peripheral Capillary Oxygen Saturation (SpO2, %) [Median (Inter-Quartile Range); unit: percent oxygen saturation] | 97 [95 to 98] | 97 [95 to 98] | 97 [95 to 98]
Systolic blood pressure (mmHg) [Median (Inter-Quartile Range); unit: mmHg] | 118 [104 to 134] | 118 [105 to 135.5] | 118 [104 to 134]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Progression to a Higher Stage of AKI OR Dialysis OR Death
Description: Progression of AKI is defined as the increase in KDIGO stage from the time of randomization to the present. For patients who are discharged, we will impute 14-day creatinine using the last observation carried forward method.
  Dialysis is defined as the receipt of hemodialysis, continuous renal replacement therapy, or peritoneal dialysis. Isolated ultrafiltration treatments will not be included.
  Mortality will be determined from hospital administrative records.
Time Frame: Within 14 days from randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Recommended | Anti-recommended
Number analyzed (Participants) | 1002 | 1044
Participants | 190 | 193

2. Secondary Outcome: 14-day Mortality
Description: Proportion of patients who expire from any cause
Time Frame: Assessed from point of randomization to date of death within 14 days of randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Recommended | Anti-recommended
Number analyzed (Participants) | 1002 | 1044
Participants | 72 | 58

3. Secondary Outcome: Inpatient Mortality
Description: Proportion of patients who expire from any cause
Time Frame: Assessed from point of randomization to date of death from any cause, up to one year post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Recommended | Anti-recommended
Number analyzed (Participants) | 1002 | 1044
Participants | 169 | 185

4. Secondary Outcome: 14-day Dialysis
Description: Proportion of patients who receive dialysis (hemodialysis, continuous renal replacement therapy, or peritoneal dialysis)
Time Frame: Assessed from point of randomization to date of first documented dialysis order, within 14 days of randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Recommended | Anti-recommended
Number analyzed (Participants) | 1002 | 1044
Participants | 38 | 37

5. Secondary Outcome: Inpatient Dialysis
Description: as for outcome 4
Time Frame: Assess from point of randomization to date of first documented dialysis order during index hospitalization, up to one year post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Recommended | Anti-recommended
Number analyzed (Participants) | 1002 | 1044
Participants | 39 | 41

6. Secondary Outcome: Discharge on Dialysis
Description: Assessed as active orders for dialysis at point of discharge from index hospitalization
Time Frame: Assessed at point of discharge from index hospitalization, up to one year post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Recommended | Anti-recommended
Number analyzed (Participants) | 1002 | 1044
Participants | 28 | 22

7. Secondary Outcome: Progression to Stage 2 AKI
Description: Progression to Stage 2 AKI is defined as a doubling of serum creatinine between randomization and 14 days post randomization, and is considered a worsening of AKI.
Time Frame: Assessed from the date of randomization to 14 days post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Recommended | Anti-recommended
Number analyzed (Participants) | 1002 | 1044
Participants | 91 | 103

8. Secondary Outcome: Progression to Stage 3 AKI
Description: Progression to Stage 3 AKI is defined as a tripling of serum creatinine between the date of randomization and 14 days post randomization, and is considered a worsening of AKI.
Time Frame: Assessed from the date of randomization to 14 days post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Recommended | Anti-recommended
Number analyzed (Participants) | 1002 | 1044
Participants | 72 | 66

9. Secondary Outcome: Duration of AKI
Description: Defined as the time in hours between AKI onset and AKI cessation during index hospitalization
Time Frame: Assessed from the date of randomization to the cessation of AKI during index hospitalization, up to one year
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Recommended | Anti-recommended
Number analyzed (Participants) | 1002 | 1044
Hours | 26.9 [22.5 to 50.1] | 27.7 [22.3 to 50.6]

10. Secondary Outcome: 30 Day Readmission Rate
Description: Proportion of patients with readmission within 30 days of index hospitalization discharge
Time Frame: Assessed from discharge date of index hospitalization to 30 days post discharge date
Measure: Count of Participants; unit: Participants
Arm/Group | Recommended | Anti-recommended
Number analyzed (Participants) | 1002 | 1044
Participants | 123 | 187

11. Secondary Outcome: Index Hospitalization Cost
Description: Total cost of index hospitalization
Time Frame: Assessed from point of randomization to date of discharge from index hospitalization, up to one year
Population: The data for this outcome were not collected and will not be accessed in the future. During outcome assessment, PIs were unable to get access to financial data to assess this outcome due to lack of institutional approval, therefore, no participants were analyzed. As this is the only financial-based outcome of the trial, this is the only outcome affected by this circumstance.
Arm/Group | Recommended | Anti-recommended
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Chart Documentation of AKI
Description: Proportion of patients with chart documentation of AKI as assessed by post-discharge ICD-10 codes
Time Frame: Assessed from date of randomization to date of discharge from index hospitalization, up to one year
Measure: Count of Participants; unit: Participants
Arm/Group | Recommended | Anti-recommended
Number analyzed (Participants) | 1002 | 1044
Participants | 442 | 505

13. Secondary Outcome: Proportion of AKI "Best Practices" Achieved Per Subject During Index Hospitalization
Description: Contrast administration (de novo order of IV contrast agent within 24 hours of randomization), fluid administration (within 24 hours of randomization), aminoglycoside administration (de novo order within 24 hours of randomization), NSAID administration/cessation (de novo order or cessation of order/absence of de novo order of NSAID within 24 hours of randomization), ACE inhibitor administration/cessation, urinalysis order (with or without microscopy within 24 hours of randomization), documentation of AKI (by ICD-9 and ICD-10 codes during index hospitalization), monitoring of creatinine (at least one serum creatinine measurement within 36 hours of randomization), documentation of urine output (within 24 hours of randomization), renal consult order during index hospitalization. Each metric is binary. Outcome is reported as a composite best practice outcome representing the proportion of best practices achieved per subject.
Time Frame: 24 hours from randomization to discharge, up to one year post randomization
Measure: Median (Inter-Quartile Range); unit: Proportion achieved per subject
Arm/Group | Recommended | Anti-recommended
Number analyzed (Participants) | 1002 | 1044
Proportion achieved per subject | .6 [.5 to .7] | .6 [.5 to .7]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the course of the enrollment period and data collection follow-up, out to one year post-randomization.
Arm/Group | Recommended | Anti-recommended
All-Cause Mortality (participants affected / at risk) | 169/1002 | 185/1044
Serious Adverse Events (participants affected / at risk) | 0/1002 | 0/1044
Other Adverse Events (participants affected / at risk) | 0/1002 | 0/1044

LIMITATIONS AND CAVEATS:
This trial was randomized at the patient level, introducing the possibility of bias towards the null. It was conducted within a single health system, limiting generalizability. The alert was largely informational with no patient-specific recommendations (not accounting for AKI heterogeneity).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-26): https://cdn.clinicaltrials.gov/large-docs/77/NCT02786277/Prot_SAP_000.pdf